CLINICAL TRIAL: NCT04838795
Title: Open-label, Single-arm Phase 3B Implementation Study to Monitor the Effectiveness of the Single-dose Ad26.COV2.S COVID-19 Vaccine Among Health Care Workers in South Africa (VAC31518COV3012)
Brief Title: Sisonke (Together): OPEN LABEL TRIAL COVID-19
Acronym: Sisonke
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wits Health Consortium (Pty) Ltd (Other)
Collaborators: National Department of Health of South Africa (Unknown); National Institute for Communicable Diseases, South Africa (Other); KwaZulu-Natal Research Innovation and Sequencing Platform - KRISP (Unknown); Fred Hutchinson Cancer Center (Other); Hutchinson Center Research Institute of South Africa (HCRISA) (Unknown); Janssen Vaccines & Prevention B.V. (Industry); Bio Analytical Research Corporation (Industry); Dis-Chem Pharmacy (Unknown); BioVac (Unknown); Biocair (Unknown); Right to Care (Other); Clinical Laboratory Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Sisonke (Together): OPEN LABEL
Record Dates: First submitted 2021-02-17; First posted 2021-04-09 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2021-10

CONDITIONS: SARS (Severe Acute Respiratory Syndrome)
MeSH Terms: conditions — Severe Acute Respiratory Syndrome

STUDY DESIGN:
Intervention Model Description: Open-label, single-arm phase 3B vaccine implementation study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: To monitor the effectiveness of the single dose Ad26.COV2.S COVID-19 vaccine — To monitor the effectiveness of the single dose Ad26.COV2.S COVID-19 vaccine among health care workers (HCW) as compared to the general unvaccinated population in South Africa

SUMMARY:
To monitor the effectiveness of the single-dose Ad26.COV2.S COVID-19 vaccine among health care workers (HCW) in South Africa

DETAILED DESCRIPTION:
Purpose To monitor the effectiveness of the single dose Ad26.COV2.S COVID-19 vaccine among health care workers (HCW) as compared to the general unvaccinated population in South Africa

Study design Open-label, single-arm phase 3B vaccine implementation study

Rationale South Africa is severely affected by the global COVID-19 epidemic, but currently no vaccine has been rolled out. The recent promising results of the 'ENSEMBLE' trial conducted by Janssen in South Africa, and the availability of a limited amount of vaccine doses, provide the rationale for a cohort study of vaccinated HCWs to inform the larger vaccine rollout.

Study participants Health Care workers age 18 and above working in the South African public and private health care sector (N=500 000) Study sites Department of Health Vaccine administration sites across South Africa supported by the Sisonke (Together) (VAC31518COV3012) trial Research Site Investigators and Study Staff

Study duration Participants will receive a single dose of vaccine at enrolment; to monitor outcomes the DATCOV surveillance system and NICD line list will be reviewed for up to 2 years post-vaccination.

A sub-cohort (approx. 850-1000 people) consisting of special sub-populations will be followed up at approx. 1, 3, 6 weeks and 6 months post vaccination. This group will also have outcomes monitored for up to a further 18 months, bringing their total follow-up duration to 2 years post-vaccination

Study products Ad26.COV2.S by Janssen administered as a single injection

Primary objectives • To assess the effectiveness of Ad26.COV2.S vaccine on severe COVID, hospitalizations and deaths in HCWs as compared with the general unvaccinated population in South Africa.

Secondary objectives • To estimate the incidence of symptomatic SARS CoV-2 infections in HCW

* To estimate vaccine uptake among HCWs in South Africa
* To monitor the genetic diversity of breakthrough SARS CoV-2 infections To monitor immunological responses (neutralising, non-neutralising antibodies and T cell responses) in HCWs with breakthrough infections
* To measure baseline SARS CoV-2 antibody testing to evaluate pre-existing immunity in up to 100 000 HCWs.
* In a subgroup of participants (approx. 850-1000 people) including representative sub-populations of interest, e.g. elderly, immune compromised:

  * To compare serum neutralization and immune responses before and after vaccination at 0, 6 weeks and up to 6 months.
  * To explore clotting parameters post vaccination at weeks 0, 1, 3.
  * To monitor for asymptomatic infection

Exploratory objectives To set up a comprehensive safety desk and establish a link between the national pharmacovigilance system to assist with monitoring safety and any unexpected adverse effects

ELIGIBILITY:
Inclusion criteria

* Age 18 and older
* Health care worker in the private or public service
* The President and Deputy President of South Africa* (The President and Deputy President of South Africa have been included in the protocol to address the issue of vaccine hesitancy. )
* Willingness and ability to comply vaccination plan and other study procedures.
* Capable of giving electronic or personal signed informed consent as described in Appendix 5, which includes compliance with the requirements in this protocol.

Inclusion criteria for the sub-cohort

* Age 18 and older
* Health care worker in the private or public service
* Willingness and ability to comply with all scheduled visits, vaccination plan, laboratory tests, and other study procedures, with follow-up at an ENSEMBLE site.
* Capable of giving electronic or personal signed informed consent as described in Appendix 5, which includes compliance with the requirements in this protocol.

Exclusion criteria

* Any significant acute or chronic medical condition, situation or circumstance that in the opinion of the PI/designee makes the participant unsuitable for participation in the study, or jeopardises the safety or rights of the participant
* Participant reports being pregnant at time of enrolment, planning conception within 3 months.
* Participants who report breastfeeding at the time of enrolment will be excluded.
* Current participation in any other research studies that would interfere with the objectives of this study. The determination of whether participation in another study would be exclusionary for a given participant will be made by the PI/designee.
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (e.g., anaphylaxis) to any component of the vaccine.
* Participants who have experienced major venous and arterial thrombosis occurring with thrombocytopenia following vaccination with any COVID-19 vaccine should not enrol in Sisonke.
* Participants with a history of heparin-induced thrombocytopenia.

Note:

• Vaccination within 14-90 days with other COVID19 or non-specific vaccines are not exclusionary but should be discussed with study PI or designee.

Conditions of interest:

We note that international reports of VITT have not identified a risk factor, nor does there appear to be any prothrombotic state that indicates a risk factor for this immune response.

Nevertheless, the Sisonke study will enrol participants with chronic history of severe clotting disorders only after consultation and approval of the study Protocol Safety Review Team (PSRT).

We have identified certain specific conditions of special interest such as:

* cerebral venous sinus thrombosis,
* antiphospholipid syndrome
* Individuals on therapeutic anticoagulants for current or previous arterial or venous thrombosis or embolism

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 477102 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Number of severe COVID, hospitalizations and deaths in HCWs as compared with the general unvaccinated population in South Africa | 24 Months
  Rates of hospitalizations and deaths among vaccinated HCWs versus general unvaccinated population

SECONDARY OUTCOMES:
The number of symptomatic SARSCoV-2 infections among vaccinated HCWs | 24 Months
  Incidence rate of SARS CoV-2 infection as indicated by self-report and validation in national laboratory records.
  Rates of severe disease in HCW who are found to be RT-PCR positive at anytime up to 2 years post vaccination
The measure of genetic diversity of breakthrough SARSCoV-2 infections | 24 months
  Genetic diversity of breakthrough infection virus as determined by whole genome sequencing. This will be recovered from national laboratories.
Monitoring for asymptomatic infection in a sub-set (10 000) of HCWs | 24 Months
  Rates of asymptomatic infection at baseline and follow up using SARS CoV-2 virus and antibody testing.
Monitor for safety and any unexpected adverse effects of the vaccine administration -pharmacovigilance | 24 Months
  Conduct Pharmacovigilance to monitor for safety and adverse events Numbers of safety events and/or unexpected adverse effects reported to the study team Monitor pregnancies and pregnancy outcomes reported to safety desk.
The vaccine uptake among HCWs in South Africa | 12 Months
  Proportion of HCWs approached for study participation taking part in the study and receiving the vaccine

OTHER OUTCOMES:
To monitor for safety and any unexpected adverse effects of the vaccine administration | 24 Months
  To conduct pharmacovigilance to monitor for safety and any unexpected adverse effects of the vaccine administration

CONTACTS AND LOCATIONS:
Overall Officials: Glenda E Gray, MBChB, Principal Investigator — Non-Executive Director
Locations (31):
- South Africa (31):
  - Nelson Mandela Academic Clinical Research Unit (NeMACRU), Mthatha, Eastern Cape
  - PHOENIX Pharma Pty Ltd, Port Elizabeth, Eastern Cape
  - Josha Research, Bloemfontein, Free State
  - CRISMO Research Centre, Dr Bhekithemba, Germiston, Gauteng
  - Perinatal HIV Research Unit (PHRU), SOWETO, Johannesburg, Gauteng
  - Wits RHI: Shandukani Research Centre, Johannesburg, Gauteng
  - Themba Lethu HIV Research Unit (CHRU), Dr, Johannesburg, Gauteng
  - Synexus SA - Stanza Clinical Research Centre, Pretoria, Gauteng
  - Setshaba Research Centre,, Pretoria, Gauteng
  - Synexus Watermeyer Clinical Research Centre,, Pretoria, Gauteng
  - Ndlovu Research Centre, Pretoria, Gauteng
  - The Aurum Institute: Tembisa Clinical Research Centre, Johannesburg, Gauteng - South
  - Perinatal HIV Research Unit Kliptown, Johannesburg, Gauteng - South
  - Botha's Hill Clinical Research Site, Bothas Hill, KwaZulu-Natal
  - CAPRISA eThekwini Clinical Research Site, Dr, Durban, KwaZulu-Natal
  - Chatsworth Clinical Research Site, Durban, KwaZulu-Natal
  - CAPRISA Vulindlela Clinical Research Site, Dr, Durban, KwaZulu-Natal
  - Qhakaza Mbokodo Research Clinic, Ladysmith, KwaZulu-Natal
  - Tongaat Clinical Research Site, Dr, Tongaat, KwaZulu-Natal
  - Mzansi Ethical Research Centre, Middleburg, Mpumalanga
  - The Aurum Institute Klerksdorp Clinical Research Centre, Klerksdorp, North West
  - FAMCRU (Family Clinical Research Unit),, Cape Town, Western Cape
  - TASK Central, Cape Town, Western Cape
  - TASK Clinical Research Centre, Cape Town, Western Cape
  - Emavundleni Research Centre, Cape Town, Western Cape
  - Khayelitsha CRS, Dr Amy Ward / Dr Graeme Meintjes, Cape Town, Western Cape
  - Desmond Tutu Health Foundation CTU J52 Old Main Building Groote SchuurHospital, Cape Town, Western Cape
  - Synexus Helderberg Clinical Research Centre, Dr Vera, Somerset West, Western Cape
  - South African Vaccine Initiative (SATVI), Dr Angelique Kany Kany, Worcester, Western Cape
  - Desmond Tutu Health Foundation - Masiphumelele Research Office, Cape Town
  - The Aurum Institute: Rustenburg Clinical Research Centre, Dr Lawrence, Rustenburg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jacobson BF, Schapkaitz E, Takalani A, Rowji PF, Louw V, Opie J, Bekker LG, Garrett N, Goga A, Reddy T, Zuma NY, Sanne I, Seocharan I, Peter J, Robinson M, Collie S, Khan A, Takuva S, Gray G. Vascular thrombosis after single dose Ad26.COV2.S vaccine in healthcare workers in South Africa: open label, single arm, phase 3B study (Sisonke study). BMJ Med. 2023 Mar 23;2(1):e000302. doi: 10.1136/bmjmed-2022-000302. eCollection 2023. PMID 37063238
- [Derived] Takuva S, Takalani A, Seocharan I, Yende-Zuma N, Reddy T, Engelbrecht I, Faesen M, Khuto K, Whyte C, Bailey V, Trivella V, Peter J, Opie J, Louw V, Rowji P, Jacobson B, Groenewald P, Dorrington RE, Laubscher R, Bradshaw D, Moultrie H, Fairall L, Sanne I, Gail-Bekker L, Gray G, Goga A, Garrett N; Sisonke study team. Safety evaluation of the single-dose Ad26.COV2.S vaccine among healthcare workers in the Sisonke study in South Africa: A phase 3b implementation trial. PLoS Med. 2022 Jun 21;19(6):e1004024. doi: 10.1371/journal.pmed.1004024. eCollection 2022 Jun. PMID 35727802
- [Derived] Bekker LG, Garrett N, Goga A, Fairall L, Reddy T, Yende-Zuma N, Kassanjee R, Collie S, Sanne I, Boulle A, Seocharan I, Engelbrecht I, Davies MA, Champion J, Chen T, Bennett S, Mametja S, Semenya M, Moultrie H, de Oliveira T, Lessells RJ, Cohen C, Jassat W, Groome M, Von Gottberg A, Le Roux E, Khuto K, Barouch D, Mahomed H, Wolmarans M, Rousseau P, Bradshaw D, Mulder M, Opie J, Louw V, Jacobson B, Rowji P, Peter JG, Takalani A, Odhiambo J, Mayat F, Takuva S, Corey L, Gray GE; Sisonke Protocol Team; Sisonke Study Team. Effectiveness of the Ad26.COV2.S vaccine in health-care workers in South Africa (the Sisonke study): results from a single-arm, open-label, phase 3B, implementation study. Lancet. 2022 Mar 19;399(10330):1141-1153. doi: 10.1016/S0140-6736(22)00007-1. PMID 35305740